CLINICAL TRIAL: NCT02003391
Title: Prospective, Randomized, Multi-Center Study to Evaluate the Efficacy and Tolerability of DuoTrav® in Patients Previously Uncontrolled on a Beta-blocker
Brief Title: Efficacy of Travoprost/Timolol for Uncontrolled Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-13-038
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular Hypertension; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DuoTrav (Experimental): Travoprost 0.004% / timolol 0.5% fixed combination ophthalmic solution, 1 drop instilled in the study eye once daily (evening) for 8 weeks.
  Interventions: Drug: Travoprost 0.004% / timolol 0.5% fixed combination ophthalmic solution
- Beta-blocker (Active Comparator): Participant's current beta-blocker monotherapy, 1 drop instilled in the study eye twice daily (morning and evening) for 4 weeks, followed by travoprost 0.004% / timolol 0.5% fixed combination ophthalmic solution, 1 drop instilled in the study eye once daily (evening) for 4 additional weeks.
  Interventions: Drug: Beta-blocker monotherapy; Drug: Travoprost 0.004% / timolol 0.5% fixed combination ophthalmic solution

INTERVENTIONS:
Drug: Beta-blocker monotherapy — Per participant's current prescribed therapy
  Arms: Beta-blocker
Drug: Travoprost 0.004% / timolol 0.5% fixed combination ophthalmic solution
  Other Names: DUOTRAV®

SUMMARY:
The purpose of this study is to demonstrate superior intraocular pressure (IOP) control with travoprost 0.004% / timolol 0.5% compared to beta-blocker monotherapy in participants with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of either open angle glaucoma or ocular hypertension.
* Currently on beta-blocker monotherapy (for >30 days) and would benefit, in the opinion of the investigator, from further intraocular pressure (lOP) reduction.
* Have a mean baseline lOP of >18 mmHg and <32 mmHg in at least one eye.
* Must be able to understand and sign an Informed Consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Use of medication excluded by the protocol.
* Diseases, illnesses, infections, or ocular abnormalities excluded by the protocol.
* Ocular surgeries or procedures excluded by the protocol.
* Best-corrected visual acuity (BCVA) score worse than 55 ETDRS letters (equivalent to 20/80 Snellen, 0.60 logMAR or 0.25 decimal).
* Hypersensitivity to prostaglandin analogues or any component of the study medications in the opinion of the investigator.
* Women of childbearing potential if pregnant, test positive for pregnancy at Screening visit, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead GCRA, Pharma, Study Director — Alcon Research

REFERENCES:
- [Derived] Lerner SF, Park KH, Hubatsch DA, Erichev V, Paczka JA, Roberts TV. Efficacy and Tolerability of Travoprost 0.004%/Timolol 0.5% Fixed-Dose Combination for the Treatment of Primary Open-Angle Glaucoma or Ocular Hypertension Inadequately Controlled with Beta-Blocker Monotherapy. J Ophthalmol. 2017;2017:1917570. doi: 10.1155/2017/1917570. Epub 2017 Jan 23. PMID 28239491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 14 investigational centers located in Latin America, Australia, Russia, and Korea.
Pre-assignment Details: Of the 157 participants enrolled, 1 participant was exited as a screen failure. This reporting group includes all randomized participants (156).
Groups:
- DuoTrav: Travoprost/timolol for 8 weeks
- Beta-blocker: 4 weeks of beta-blocker monotherapy, followed by 4 weeks of travoprost/timolol
Period: Overall Study
Arm/Group | DuoTrav | Beta-blocker
Started | 81 | 75
Safety Population | 81 | 75
Intent to Treat Population | 78 | 73
Completed | 78 | 73
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population included participants who received study medication and had at least one on-therapy study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | DuoTrav | Beta-blocker | Total
Number analyzed (Participants) | 78 | 73 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (12.76) | 63.8 (13.29) | 63.3 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Intraocular Pressure (IOP) at 8AM in the Study Eye
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and is measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) contributed to the analysis.
Time Frame: Week 4
Population: Intent to treat with a measurement in the study eye at Week 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- DuoTrav: Travoprost/timolol for 4 weeks
- Beta-blocker: Beta-blocker monotherapy for 4 weeks
Arm/Group | DuoTrav | Beta-blocker
Number analyzed (Participants) | 78 | 72
mmHg | 16.6129 [NA to 17.1451] — NA = not quantifiable (calculated to infinity) | 21.2320 [NA to 21.7858] — NA = not quantifiable (calculated to infinity)
Statistical Analysis 1: Comparison: DuoTrav vs Beta-blocker; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.6191, 95% CI 1-sided [upper limit -3.8503]

2. Secondary Outcome: Mean Change From Baseline in IOP (8AM) at Week 4 in the Study Eye
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and is measured in mmHg. A negative change indicates an improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Intent to treat with a measurement in the study eye at Week 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DuoTrav | Beta-blocker
Number analyzed (Participants) | 78 | 72
mmHg | -5.840 (3.4870) | -1.069 (2.4969)

3. Secondary Outcome: Percentage Change From Baseline in IOP (8AM) at Week 4 in the Study Eye
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and is measured in mmHg. A more negative percent change from baseline indicates a greater amount of improvement, i.e., a reduction of IOP. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Intent to treat with a measurement in the study eye at Week 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | DuoTrav | Beta-blocker
Number analyzed (Participants) | 78 | 72
Percent Change | -25.365 (14.2093) | -4.716 (11.4005)

ADVERSE EVENTS:
Time Frame: Reporting of adverse events (AEs) began once informed consent was obtained from the participant and continued through study exit at week 8. Ocular AEs are presented for both study eye and non-study eye combined.
Description: An AE was defined as any untoward medical occurrence in a participant who was administered study treatment regardless of whether or not the event had a causal relationship to study treatment. AEs were reported as pre-treatment and treatment-emergent. Reports of AEs were obtained through solicited and spontaneous comments from the participants.
Arm/Group | DuoTrav | Beta-blocker
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/75
Other Adverse Events (participants affected / at risk) | 18/81 | 9/75
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DuoTrav (N=81) | Beta-blocker (N=75)
Blepharal pigmentation (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 2 | 2
Eye irritation (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 4 | 0
Eyelids pruritus (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 5 | 0
Ocular surface disease (Eye disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.